CLINICAL TRIAL: NCT06690814
Title: Ulcer Plants: Highly Accessible Plant Antiseptics for Use in Remote Areas of PNG
Acronym: UP2024
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: The Royal Botanic Gardens, Kew (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UlcerPlants2024
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Ulcer Disease; Skin Sores
Keywords: sap; cutaneous ulcers; plant sap; antiseptic plant; papua new guinea; infected skin sores
MeSH Terms: conditions — Skin Ulcer; Lymphoproliferative Disorders | interventions — Cetrimonium; chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: The study we propose is an evaluator-blinded, randomized clinical trial to compare the effects of topical application of three traditional medicine plant saps compared to Savlon cream or no treatment:
  (A) Ficus septica plant sap (50μl) applied topically at baseline, day 3 and day 7.
  (B) Pterocarpus indicus plant sap (50μl) applied topically at baseline, day 3 and day 7.
  (C) Curcuma longa plant sap (50μl) applied topically at baseline, day 3 and day 7.
  (D) Savlon cream (200mg) applied topically at baseline, day 3 and day 7. (E) No treatment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Ficus septica exudate (Experimental)
  Interventions: Other: Ficus septica exudate (antiseptic plant exudates)
- Pterocarpus indicus exudate (Experimental)
  Interventions: Other: Pterocarpus indicus exudate
- Curcuma longa aqueous extract (Experimental)
  Interventions: Other: Curcuma longa aqueous extract
- Savlon antiseptic cream (cetrimide with chlorhexidine digluconate ) (Active Comparator)
  Interventions: Drug: Savlon antiseptic cream (cetrimide with chlorhexidine digluconate)
- Control (No Intervention)

INTERVENTIONS:
Other: Ficus septica exudate (antiseptic plant exudates) — F. septica sap contains the antibacterial alkaloid ficuseptine which exhibits activivity agaisnt S. pyogenes and H. ducreyi, two pàthogens associated with cutaneous ulcer disease in Papau New Guinea. The sap has been tested using the Ames test for mutagenesis, and found to be non-mutagenic; testing was carried out by toxicology service provider Gentronix, UK (results available separately on request).
  Arms: Ficus septica exudate
Other: Pterocarpus indicus exudate — P. indicus sap exhibits antibacterial activivity agaisnt S. pyogenes, a pàthogen associated with cutaneous ulcer disease in Papau New Guinea. The sap has been tested using the Ames test for mutagenesis, and found to be non-mutagenic; testing was carried out by toxicology service provider Gentronix, UK (results available separately on request).
  Arms: Pterocarpus indicus exudate
Other: Curcuma longa aqueous extract — C. longa is a culinary herb that contains the antibatieral compound curcumin. Curcumin exhibits antibacterial activity agasint S. pyogenes and has profound effects on bacterial biofilms. This intervention uses a mulch of the rhizome that has been sqeeezed to produce a curcumin containing aqueous fluid.
  Arms: Curcuma longa aqueous extract
Drug: Savlon antiseptic cream (cetrimide with chlorhexidine digluconate) — Common over the counter antiseptic cream
  Arms: Savlon antiseptic cream (cetrimide with chlorhexidine digluconate )

SUMMARY:
Small cutaneous ulcers are common in Papua New Guinea but are normally left untreated due to lack of easy access to basic medicines. The goal of this clinical trial is to test the efficacy of three readily available antibacterial plant medicines, Ficus septica, Pterocarpus indicus and Curcuma longa, comparing healing outcomes to control arms receiving Savlon antiseptic cream or no treatment. Participants with cutaneous ulcers less than 1cm in diameter will be randomized to receive topical treatment with one of three different plant medicines, Savlon cream or no treatment treatment and followed up at day 7 and 14 to assess ulcer healing and ulcer surface area.

DETAILED DESCRIPTION:
Small, infected skin ulcers are very common in children living in rural areas of Papua New Guinea (PNG) and represent a large area of unmet clinical need. These painful and debilitating ulcers often occur on the lower leg area and are suspected to be associated with a range of different bacterial pathogens including Haemophilus ducreyi and Streptococcus pyogenes. Topical antiseptics such as chlorhexidine-based antiseptic creams or antibiotics such as amoxicillin may be effective treatment options, but in rural areas of PNG, infected skin ulcers are normally left untreated due to a lack of access to such treatments. The need to walk many miles to reach an aid post, often barefoot and through swampy or muddy ground, compromises the real-world effectiveness of such treatments in PNG. In this study we propose to test the effectiveness of three antibacterial traditional plant medicines, each of which has a long history of use in PNG as a plant-based topical antiseptic that is applied directly onto infected skin ulcers. The three plant medicines Ficus septica, Pterocarpus indicus and Curcuma longa each comprise antibacterial plant saps which as viscous fluids can be easily applied directly onto the surface of infected ulcers. Unlike antibiotics such as amoxicillin which demand access to an aid post or clinic, these plant medicines can be easily found growing in or very near to most villages in PNG. Highly accessible, medicinal plant saps could form the basis of a cost-effective treatment option for PNG in remote areas, and may reduce the use of antibiotics. The trial proposed in this application aims to discover if such plant medicines are indeed efficacious when compared to Savlon cream or no treatment.

The aim of the project is to provide evidence supporting or rejecting the hypothesis that the use of one of more of these antibacterial plant medicines can improve healing or reduce the severity of small cutaneous ulcers in Papua New Guinea. Participants with ulcers less than 1cm in largest diameter will be recruited and randomised into one of five treatment arms, images and dimensions of ulcers will be recorded at baseline. Participants will receive topical treatment with one of the three plant saps, Savlon antiseptic cream or will receive no treatment. Investigators will compare healing and size of ulcers at day 7 and day 14. The study will be implemented in selected wards of East New Britain Province in Papua New Guinea.

ELIGIBILITY:
Inclusion Criteria:

* Infected skin ulcer suspected with one or more predominantly moist ulcerative skin lesions of less than 1 cm diameter in greatest dimension and larger than 0.5cm in largest dimension with a predominantly moist surface, occurring below the knee.
* Accepted and signed informed consent by a legal guardian (relative or teacher)
* Ability and willingness to comply with the requirements of the study protocol including follow up visits.

Exclusion Criteria:

* Children younger than 5 years old.
* Ulcer presenting with a crust (not predominantly moist surface), or dimensions different to those specified in point 1 above.
* Refusal at ward level or village chief (for village inclusion), or refusal of individual or guardian (for individual inclusion).
* Answered yes when asked if had taken antibiotics in the last week or presents with visible signs of ulcer treatment e.g. wound dressing.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 370 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Wound healing | 2 weeks
  A wound diameter reduction of more than 25% measured by the eKare wound imaging system.

CONTACTS AND LOCATIONS:
Locations (1):
- Vunapope Hospital, Kokopo, EAST NEW Britan, Papua New Guinea

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request within a reasonable time-frame.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 months